CLINICAL TRIAL: NCT04245813
Title: Effectiveness of a Cardiac Rehabilitation Program in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Rehabilitacion en Salud (Network)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Universidad de Antioquia (Other); Clinica Las Americas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111580763152
Record Dates: First submitted 2019-12-17; First posted 2020-01-29 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Consists of 3 interdisciplinary educational sessions and Face-to-face with a fortnightly telephone follow-up and text messages. Each session will be directed by medical staff (cardiologist and / or physiatrist) and supported by other health professionals (physical therapist, occupational therapist, nutritionist and psychologist). The educational sessions, include the topics "knowledge of the disease", "recognition of alarm signs", "pharmacological treatment", "healthy lifestyle habits", "mental health" and "regular aerobic exercise"; The entire educational component will be based on the Colombian clinical practice guide for the prevention, diagnosis, treatment and rehabilitation of heart failure.
  Interventions: Behavioral: Interdisciplinary educational program
- Control (No Intervention): Once the patient ends phase II of the cardiac rehabilitation program, he/she will receive the usual care, which consists of a 5-minute educational intervention by a physiatrist at the end of the functional test, where recommendations are given on healthy lifestyle habits, adherence to pharmacological treatment and regular aerobic exercise. This educational intervention will be performed after each of the functional tests (at the end of phase II of the program and during the follow-up of patients at months 1, 3, 6 and 12 during Phase III of the program) performing 5 educational interventions in total .

INTERVENTIONS:
Behavioral: Interdisciplinary educational program — Interdisciplinary educational component based on the Clinical Practice Guide for Heart Failure
  Arms: Intervention

SUMMARY:
Heart failure is a devastating disease with great impact on the quality of life and survival of those who suffer from it. The disease has a high prevalence and its treatment represents high economic costs for health systems. In Colombia, cardiovascular diseases that are part of chronic noncommunicable diseases are the first cause of death. According to figures from the World Health Organization (WHO) in 2014, 28% of deaths in the country were due to cardiovascular diseases.

Pharmacological treatment, patient education and regular physical activity are the cornerstones for the treatment of heart failure and therefore the international clinical practice guidelines as well as the guide of the Colombian Ministry of Health recommend the performance of supervised physical exercise for patients with the disease. Cardiac rehabilitation programs using regular and supervised aerobic exercise positively impact the lives of these patients by improving functional capacity, quality of life, psychological well-being and can have an effect on important outcomes. such as hospitalizations and mortality.

The Health Rehabilitation Group has carried out several research projects on heart failure and other cardiovascular diseases, and in agreement with the Ministry of Health and Social Protection (COLCIENCIAS) developed the Clinical Practice Guide for the Prevention, Diagnosis, Treatment and Rehabilitation of Heart Failure in population over 18 years of age classification B, C and D. The group's research has demonstrated the efficacy and safety of cardiac rehabilitation to improve functional capacity, abdominal perimeter and systemic blood pressure figures in patients with cardiovascular diseases, improvement in the quality of life in patients with heart failure and the prevalence of musculoskeletal diseases has even been described in this group of patients. In one of the studies, an exercise program was compared with an educational program and it was concluded that the exercise was effective in improving the health-related quality of life of patients with heart failure.

Despite the benefits demonstrated by the cardiac rehabilitation programs, the adherence to exercise of the patients is low, especially during phase III of the program in which patients exercise in an unsupervised manner with periodic care follow-up. In some studies they have carried out other types of follow-up such as telephone control, home visits and telemonitoring, but there are no studies that carry out a low-cost program, with telephone follow-up and distance education to improve adherence in the phase III of cardiac rehabilitation.

The aim of this study is to determine the effect of an education, follow-up and stimulus program of adherence to the achievements of phase III of the Rehabilitation Program in patients with heart failure, on functional capacity, quality of life, the need to return to phase II of the program and rehospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Spanish language.
* Live in Medellin or near the city municipalities.
* Available to attend the face-up meetings.
* Accepts to participate in the study.
* Have completed Phase II cardiac rehabilitation.
* Have a confirmed diagnosis of heart failure with ejection fraction measured by echocardiography, scintigraphy or cardiac resonance. For cases with expulsion fraction> 40%, it is required to have high levels of natriuretic peptides.
* New York Heart Association (NYHA) functional class II and III.

Exclusion Criteria:

* Acute coronary syndrome not treated in the last month.
* Severe symptomatic aortic stenosis.
* Atrial fibrillation with uncontrolled ventricular response.
* Symptomatic or hemodynamic compromise cardiac arrhythmias.
* New York Heart Association (NYHA) functional class IV or that requires the use of parenteral medications such as diuretics or inotropics (in-hospital or outpatient).
* Myocarditis or acute pericarditis.
* Previous aortic dissection.
* Poorly controlled systemic arterial hypertension.
* Recent pulmonary thromboembolism.
* Chronic obstructive pulmonary disease.
* Restrictive lung disease.
* Osteomuscular disease that limits physical activity.
* Cognitive and / or behavioral disorders that prevent the understanding of instructions.
* Difficulty in developing questionnaires in Spanish due to cultural differences.
* Diabetes mellitus decompensated.
* Be participating in another clinical trial.
* Participants who previously did NOT complete the cardiac rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to the program in one year (Questionnaire) | One year
  The proportion of adherent patients will be estimated one year after the end of phase II of cardiac rehabilitation in each arm of the study and the relative risk will be calculated with their respective 95% confidence interval.

SECONDARY OUTCOMES:
Adherence to the program at 1, 3 and 6 months (Questionnaire) | Months 1, 3 and 6
  The proportion of adherent patients will be estimated in each of the periods followed (1, 3 and 6 months) after the end of phase II of cardiac rehabilitation in each arm of the study. The relative risk will be calculated with its respective 95% confidence interval for each of the periods.
Functional performance (Stress test with exercise) | Months 1, 3, 6 and 12
  Stress test
Minnesota Living with heart Failure Questionnaire and The Duke Activity Status Index (DASI) | Months 1, 3, 6 and 12
  Minnesota Living with heart Failure Questionnaire and The Duke Activity Status Index (DASI)
Return to phase II of rehabilitation | Months 1, 3, 6 and 12
  Return to phase II of rehabilitation
Hospitalizations | Months 1, 3, 6 and 12
  Hospitalizations due to cardiac disease
Death | Months 1, 3, 6 and 12
  Death of cardiac diseases or other causes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica de Las Américas, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No